CLINICAL TRIAL: NCT04920617
Title: A Phase 2b, Open-label, Multicenter, Randomized Parallel-Group, Two-Stage, Study of an Immunotherapeutic Treatment DPX-Survivac and Pembrolizumab, With and Without Intermittent Low-Dose Cyclophosphamide, in Subjects With Relapsed/Refractory Diffuse Large B-Cell Lymphoma (VITALIZE)
Brief Title: DPX-Survivac and Pembrolizumab With and Without Intermittent Low-Dose Cyclophosphamide, in Subjects With Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Acronym: VITALIZE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ImmunoVaccine Technologies, Inc. (IMV Inc.) (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1605-SUR-D23; KEYNOTE-C54 (Other: Merck Sharp & Dohme Corp.)
Record Dates: First submitted 2021-05-28; First posted 2021-06-10 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2022-08

CONDITIONS: Relapsed Diffuse Large B-cell Lymphoma; Refractory Diffuse Large B-cell Lymphoma
Keywords: Immunotherapy; T cell activation; DLBCL; Anti-PD-1; CAR-T ineligible; ASCT ineligible
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — pembrolizumab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: DPX-Survivac, pembrolizumab, CPA (Experimental): Subjects will receive two 0.5 mL doses of DPX-Survivac three weeks apart followed by up to twelve 0.1 mL doses eight weeks apart. Pembrolizumab will be administered on the first day of every three week cycle at a flat dose of 200 mg. CPA will be self-administered 50 mg BID for 7 days on and 7 days off starting on D0.
  Interventions: Drug: DPX-Survivac; Drug: Pembrolizumab; Drug: CPA
- Arm 2: DPX-Survivac, pembrolizumab (Experimental): Subjects will receive two 0.5 mL doses of DPX-Survivac three weeks apart followed by up to twelve 0.1 mL doses eight weeks apart. Pembrolizumab will be administered on the first day of every three week cycle at a flat dose of 200 mg. Subjects randomized to Arm 2 will not receive CPA.
  Interventions: Drug: DPX-Survivac; Drug: Pembrolizumab

INTERVENTIONS:
Drug: DPX-Survivac — SC injection on D7 and D28, then every 8 weeks
  Other Names: maveropepimut-S
Drug: Pembrolizumab — IV infusion every 3 weeks
  Other Names: MK-3475; Keytruda
Drug: CPA — 50 mg twice daily, week on then week off
  Other Names: Intermittent, low-dose cyclophosphamide; Procytox; Cytoxan
  Arms: Arm 1: DPX-Survivac, pembrolizumab, CPA

SUMMARY:
This is a Phase 2b, randomized, open label study to assess the safety and efficacy of DPX-Survivac and pembrolizumab, with and without low-dose cyclophosphamide (CPA) in subjects with relapsed or refractory DLBCL.

DETAILED DESCRIPTION:
This is a Phase 2b, randomized, open label study to assess the safety and efficacy of DPX-Survivac and pembrolizumab, with and without low-dose cyclophosphamide (CPA) in subjects with relapsed or refractory DLBCL.

The study will enroll up to 102 subjects. Eligible subjects will be randomized (1:1) to receive:

* Arm 1: DPX-Survivac, pembrolizumab and intermittent, low-dose CPA; or,
* Arm 2: DPX-Survivac and pembrolizumab

All subjects will receive two 0.5 mL doses of DPX-Survivac 3 weeks apart on day 7 (D7) and D28 followed by up to twelve 0.1 mL doses of DPX-Survivac, 8 weeks apart (Q8W).

All subjects will receive pembrolizumab intravenously (IV) at a flat dose of 200 mg starting at D7 and on day 1 of each 3-week cycle thereafter (i.e., D28, D49, D70 etc.) (Q3W).

For subjects randomized to Arm 1, intermittent oral CPA at a dose of 50 mg twice a day (BID) is administered from D0 to D6 (7 days) followed by 7 days off. This 14-day cycle of "7 days on and 7 days off" will be repeated until the end of study treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Adults ≥ 18 years of age who are willing and able to provide written informed consent
* Have an ECOG performance status of ≤ 1. Subjects with an ECOG performance status of 2 may be enrolled with Medical Monitor approval.
* Pathologically confirmed diagnosis of DLBCL, as defined by the 2016 World Health Organization classification including DLBCL NOS high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements, Epstein-barr virus (EBV) positive DLBCL, and T cell rich B cell lymphoma (TCRBCL). Subjects with DLBCL transformed from indolent lymphoma (except for Richter's transformation) are eligible.
* Subjects must have progressive disease following at least two (2) lines of prior systemic therapy for DLBCL; prior treatment must have included an anthracycline and rituximab (or another CD20-targeted agent).
* Subjects must have failed or be ineligible for ASCT or CAR-T
* Have at least one bi-dimensionally measurable lesion per Lugano (2014)
* Willing to provide pre-treatment and on-treatment tumor biopsy tissue.
* Meet protocol-specified laboratory requirements
* Life expectancy > 3 months.

Key Exclusion Criteria:

* Primary CNS lymphoma or active secondary CNS involvement and/or lymphomatous meningitis
* Chemotherapy, immunotherapy, major surgery, or investigational agent treatment within 28 days of D0 or 5 half-lives, whichever is shorter
* Radiotherapy within 14 days of day 0
* Autologous stem cell transplant (ASCT) within ˂100 days prior to D0
* Chimeric antigen receptor T cell (CAR-T) therapy within ˂28 days prior to D0
* Diagnosis of immunodeficiency disorder or history of active autoimmune disease that has required systemic treatment in the past 2 years
* Uncontrolled significant active infections (controlled Hepatitis B, Hepatitis C, or HIV may be eligible)
* Prior history of malignancy other than eligible lymphoma sub-types, unless the subject has been free of the disease for ≥ 2 years prior to the start of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) in each of the study arms | Approximately 24 months
  Centrally evaluated using Lugano (2014)

SECONDARY OUTCOMES:
Rate of Adverse Events using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 in each of the study arms | Approximately 24 months
Duration of response (DOR) in each of the study arms | Approximately 24 months
  Centrally evaluated using Lugano (2014)
Time to response in each of the study arms | Approximately 24 months
  Centrally evaluated using Lugano (2014)
Progression-Free Survival in each of the study arms | Approximately 48 months
  Centrally evaluated using Lugano (2014)
Disease control rate (DCR) in each of the study arms | Approximately 24 months
  Centrally evaluated using Lugano (2014)
Complete response (CR) rate in each of the study arms | Approximately 24 months
  Centrally evaluated using Lugano (2014)
Changes in Patient Reported Outcomes using the FACT-Lym Assessment | Approximately 24 months
  The FACT-Lym is a validated questionnaire that consists of a 27-item general core questionnaire (i.e., Functional Assessment of Cancer Therapy - General [FACT-G]) and a 15-item disease-specific questionnaire (Lymphoma Subscale).
Changes in Patient Reported Outcomes using the EQ-5D-5L Assessment | Approximately 24 months
  The EQ-5D-5L is a 5-item measure that can be used to describe and value current overall health consisting of 5 items assessing mobility, self care, usual activities, pain/discomfort, and anxiety/depression.

OTHER OUTCOMES:
Objective Response Rate (ORR) based on PD-L1 expression | Approximately 24 months
  Centrally evaluated using Lugano (2014) and central assessment of PD-L1 using validated 22C3 assay
Time to next treatment (TTNT) in each of the study arms | Approximately 48 months
Overall survival (OS) in each of the study arms | Approximately 48 months
Time to second objective disease progression (PFS2) in each of the study arms | Approximately 48 months
Cell mediated immune response | Approximately 24 months
Changes in immune cell infiltration in tumor biopsies | Approximately 24 months

CONTACTS AND LOCATIONS:
Locations (50):
- United States (17):
  - Compassionate Cancer Care Medical Group, Fountain Valley, California
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - BRCR Medical Center Inc., Hollywood, Florida
  - BRCR Medical Center Inc., Plantation, Florida
  - Comprehensive Hematology and Oncology, St. Petersburg, Florida
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Tulane Cancer Center Office of Clinical Research, New Orleans, Louisiana
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Christus St. Vincent Regional Cancer Center, Santa Fe, New Mexico
  - Brody School of Medicine at East Carolina University, Greenville, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - Allegheny Health Network (AHN) West Penn Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital - McGlinn Cancer Institute, West Reading, Pennsylvania
  - Prairie Lakes Health Care System, Watertown, South Dakota
- Australia (4):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Epworth Freemasons Hospital, Melbourne, Victoria
  - Box Hill Hospital, Melbourne, Victoria
  - Westmead Hospital, Westmead
- Saskatoon Cancer Center, Saskatoon, Saskatchewan, Canada
- France (10):
  - Hôpital Avicenne, Bobigny
  - Centre d'Oncologie de Gentilly, Nancy
  - Hôpital Privé du Confluent, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hôpital Saint-Antoine, Paris
  - Hôpital de la Pitié-Salpêtrière, Paris
  - Hôpital Necker, Paris
  - CHU Bordeaux- Hôpital Haut Lévêque, Pessac
  - Centre Hospitalier de Périgueux, Périgueux
  - Centre Hospitalier de Saint-Quentin, Saint-Quentin
- Hungary (2):
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - SzSzBM Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
- New Zealand (2):
  - North Shore Hospital, Auckland, Auckland Province
  - Palmerston North Hospital, Palmerston North, Manawatu
- Poland (5):
  - Szpitale Pomorskie Sp. z o. o., Gdynia
  - Wojewódzki Szpital Specjalistyczny w Legnicy, Legnica
  - SP ZOZ MSWiA z Warmińsko-Mazurskim Centrum Onkologii w Olsztynie, Olsztyn
  - Centrum Medyczne Pratia Poznań, Skórzewo
  - Narodowy Instytut Onkologii im. Marii, Skłodowskiej-Curie, Warsaw
- Romania (2):
  - Bucharest Oncology Institute "Prof.Dr.Al. Trestioreanu", Bucharest
  - The Oncology Institute "Prof. Dr. Ion Chiricuţă" I.O.C.H., Cluj-Napoca
- Serbia (4):
  - University Clinical Center of Serbia, Belgrade
  - Oncology Institute of Vojvodina, Kamenitz
  - University Clinical Center Kragujevac, Kragujevac
  - Clinical Hospital Center Zemun, Zemun
- Spain (3):
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Virgen del Rocío, Seville